CLINICAL TRIAL: NCT00887627
Title: A Phase 1, Open-Label Study to Assess the Effects of Renal Impairment on the Pharmacokinetics of Intravenous Conivaptan
Brief Title: Study to Compare Conivaptan Pharmacokinetics in Subjects With Mild & Moderate Kidney Function Impairment to Subjects With Normal Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 087-CL-094
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Kidney Diseases; Hyponatremia
Keywords: Pharmacokinetics; Protein Binding; Conivaptan; Vaprisol; Kidney Diseases
MeSH Terms: conditions — Kidney Diseases; Hyponatremia | interventions — conivaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1. Mild Renal Function Impaired Subjects (Experimental)
  Interventions: Drug: conivaptan hydrochloride
- 2. Moderate Renal Function Impaired Subjects (Experimental)
  Interventions: Drug: conivaptan hydrochloride
- 3. Subjects with Normal Renal Function (Experimental)
  Interventions: Drug: conivaptan hydrochloride

INTERVENTIONS:
Drug: conivaptan hydrochloride — intravenous
  Other Names: Vaprisol; YM087

SUMMARY:
A study to compare a conivaptan PK in subjects with mild or moderate kidney function impairment to subjects with normal kidney function after a 48-hour continuous infusion of conivaptan.

ELIGIBILITY:
Inclusion Criteria:

* Weighs at least 45 kg
* Body mass index between 18 and 40 kg/m2 inclusive
* Must be in good health other than renal function impairment and related stable diseases for the renal impaired subjects
* Must have a screening and pre-dose estimated glomerular filtration rate (GFR) that corresponds with the level of renal impairment based on the abbreviated Modification of Diet in Renal Disease (MDRD) formula
* Female subject of child-bearing potential must not be pregnant or lactating, must have a negative pregnancy test, utilizes adequate contraceptive methods while in this study or may be surgically sterile and/or two years post menopausal

Exclusion Criteria:

* Subject is known to be HIV positive or has HIV antibodies
* Has clinically significant history or presence of illness, medical condition, or laboratory abnormality
* Is Hepatitis positive
* Subject with renal impairment has not been on a stable dose of concomitant medications for at least 4 weeks prior to start of study and/or dose changes are likely during the study
* History of substance abuse within 6 months prior to screening
* Has clinically significant history or presence of psychiatric illness, malignancy, or immunodeficiency syndrome
* Has abnormal liver function tests (ALT, AST, and/or bilirubin)
* Has had a blood transfusion or donated/lost more than 450ml of blood within 56 days of study drug administration or has donated plasma within 7 days prior to study drug administration

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Measure PK and protein binding of conivaptan | 5 days

SECONDARY OUTCOMES:
Measure safety and tolerability of conivaptan | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Art Wheeler, MD, Study Director — Cumberland Pharmaceuticals, Inc.
Locations (1):
- Anaheim, California, United States